CLINICAL TRIAL: NCT06001502
Title: The Effect of Virtual Reality on Postoperative Pain and Anxiety in Cardiac Surgery.
Acronym: VRECOVERY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Jolanda Kluin, Professor dr. J. Kluin, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL79616.018.21
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Post Operative Pain; Post Operative Anxiety; Heart Surgery; Coronary Artery Bypass Grafting; Virtual Reality
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality group (Experimental): Virtual Reality distraction therapy on post-operative days 1,2 and 3.
  Interventions: Device: Virtual Reality distraction therapy
- Control Group (No Intervention): Conventional post-operative pain and anxiety management

INTERVENTIONS:
Device: Virtual Reality distraction therapy — The VR device simulates a 3-dimensional virtual enviroment, seeking to immerse the user in virtual surroundings
  Other Names: Healthy Mind VR device
  Arms: Virtual Reality group

SUMMARY:
The objective of this study is to investigate the effect of VR on post-operative pain and anxiety management in cardiac surgery patients undergoing a coronary artery bypass grafting (CABG) procedure.

Participants in the intervention group will receive a 20 minute session with the head mounted VR device on post-operative days 1,2 and 3.

Participants in the control group will be treated with conventional post-operative care.

DETAILED DESCRIPTION:
Objective: The objective of this study is to investigate the effect of VR on post-operative pain and anxiety management in cardiac surgery patients undergoing a coronary artery bypass grafting (CABG) procedure.

Study design: This study is a single-center randomized control trial.

Study population: Patients who have undergone a CABG procedure (n=100).

Intervention: The intervention group (n=50) will use the VR distraction therapy device at day 1, 2 and 3 after surgery on the general ward. The control group (n=50) will be treated with conventional post-operative pain and anxiety management.

Main study parameters/endpoints: The main study parameters at day 1, 2 and 3 after surgery. These are the Numeric Rating Scale (NRS) to assess the effect of pain on mobility, the Quality of Recovery-15 questionnaire, the State-Trait Anxiety Inventory-6 questionnaire and assessment of analgesic use. At follow-up, participants will be called to gather one-time QoR-15 and STAI-6 questionnaire data 6 weeks after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years or older with written informed consent
* Patients undergoing surgical CABG

Exclusion Criteria:

* Major comorbidities besides coronary artery disease
* Complicated surgical procedure
* Hearing and/or visual impairments
* Psychiatric impairments
* Complaints of vomiting and nausea
* History of epilepsy
* Claustrophobia
* Facial wounds and skin defects at site of application
* Patients placed in clinical isolation
* Readmission to the intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | Post-operative days 1,2 and 3 directly after the VR intervention
  The NRS score is a numeric scale in which individuals rate pain from 0 (no pain) tot 10 (worst pain). This is a subjective score which is assessed verbally and used frequently in standard clinical care in multiple medical specialties.
State- Trait Anxiety Inventory 6 questionnaire | Post-operative days 1,2 and 3 directly after the VR intervention
  The STAI-6 questionnaire is a validated psychological inventory designed to measure worry, tension and anxiety in an individual. It is a shortend version of the STAI score
Quality of Recovery-15 | Post-operative days 1,2 and 3 directly after the VR intervention
  The QoR-15 questionnaire is a clinical validated instrument to measure post-operative quality of recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Jolanda Kluin, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Upon request available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication
Access Criteria: Upon request available.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT06001502/Prot_SAP_000.pdf